CLINICAL TRIAL: NCT00962429
Title: Lipoic Acid for Chronic Inflammatory Demyelinating Polyneuropathy-A Randomized, Double-Blind, Placebo Controlled Pilot Study
Brief Title: Lipoic Acid to Treat Chronic Inflammatory Demyelinating Polyneuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Collins Medical Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMT-Lou
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Results first posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: CIDP; Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: neuropathy, lipoic acid
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Thioctic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lipoic acid (Active Comparator): alpha lipoic acid
  Interventions: Drug: lipoic acid
- Placebo (Placebo Comparator): sugar pill
  Interventions: Drug: lipoic acid

INTERVENTIONS:
Drug: lipoic acid — Subjects will be started on a single daily dose of 600 mg of alpha lipoic acid or placebo for the first 4 weeks and then increased to 1200 mg for the remainder of the study.
  Other Names: LA

SUMMARY:
The purpose of the study is to examine if alpha lipoic acid is an effective treatment for chronic inflammatory demyelinating polyneuropathy (CIDP).

DETAILED DESCRIPTION:
Chronic inflammatory demyelinating polyneuropathy (CIDP) is a progressive disease leading to paralysis. CIDP is an immune-mediated disorder resulting from a synergistic interaction of T cell-mediated and B cell-mediated immune responses directed against peripheral nerve antigens. These immune mediated responses in turn increase the production of reactive oxygen intermediate and cause oxidative damage of the peripheral nerve system. Although corticosteroids, plasma exchange, and intravenous immunoglobulin (IVIg) reduce impairment caused by CIDP at least temporarily and can be used as a first-line treatments, they are not ideal for long-term treatment because of serious side effects and cost. Alpha lipoic acid (LA) is an antioxidant that also possesses anti-immune activity. It is effective in treating diabetic neuropathy. It is also promising in treating patients with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CIDP
* on a stable dose of immunotherapy for at least 3 months before enrolling in the study

Exclusion Criteria:

* myelopathy or evidence of central demyelination
* persistent neurological deficits from stroke, CNS trauma, or peripheral neuropathy from other causes (eg, diabetes mellitus, IgM, paraproteinaemia, or uraemic, toxic, or familial neuropathy)
* evidence of systemic disease that might cause neuropathy
* heart diseases (congestive heart failure or arrhythmia)
* pulmonary conditions (asthma or CIPD)
* rheumatoid conditions (such as rheumatoid arthritis)
* renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Shin Lou, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Responsible Party has left the institution and has indicated that they do not have the raw data. They have confirmed that, despite all efforts to locate the data by contacting study team members, efforts were unsuccessful and no data are available.
Period: Overall Study
Arm/Group | Lipoic Acid | Placebo
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Responsible Party has left the institution and has indicated that they do not have the raw data. They have confirmed that, despite all efforts to locate the data by contacting study team members, efforts were unsuccessful and no data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lipoic Acid | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Muscle Strength
Time Frame: 16 weeks
Population: as for baseline characteristics
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Hughes Functional Disability Scale
Time Frame: 16 weeks
Population: as for baseline characteristics
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Forced Vital Capacity (FVC)
Time Frame: 16 weeks
Population: as for baseline characteristics
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Motor Nerve Conduction Studies (NCS)
Time Frame: 16 weeks
Population: as for baseline characteristics
Arm/Group | Lipoic Acid | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The Responsible Party has left the institution and has indicated that they do not have the raw data. They have confirmed that, despite all efforts to locate the data by contacting study team members, efforts were unsuccessful and no data are available.
Arm/Group | Lipoic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The Responsible Party has left the institution and has indicated that they do not have the raw data. They've confirmed that, despite all efforts to locate the data by contacting study team members, efforts were unsuccessful and no data are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes